CLINICAL TRIAL: NCT00128492
Title: A Phase 3, Open-label, Follow-On Study of Multiple Courses of Aztreonam Lysinate for Inhalation (AI) in Cystic Fibrosis Patients (AIR-CF3)
Brief Title: Safety and Efficacy Study of Aztreonam for Inhalation Solution (AZLI) in Cystic Fibrosis (CF) Patients With Pseudomonas Aeruginosa (PA)
Acronym: AIR-CF3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Mark Bresnik, MD, Director, Clinical Research, Gilead Sciences, Inc.
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CP-AI-006
Record Dates: First submitted 2005-08-08; First posted 2005-08-10 (Estimated); Results first posted 2011-03-11 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2011-05

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis; Pseudomonas aeruginosa
MeSH Terms: conditions — Cystic Fibrosis; Pseudomonas Infections | interventions — BID protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: AZLI 75 mg two times a day (BID)/ three times a day (TID)

SUMMARY:
The purpose of this study was to evaluate the safety and efficacy of multiple courses of AZLI in patients with cystic fibrosis (CF) and lung infection due to Pseudomonas aeruginosa (PA).

DETAILED DESCRIPTION:
People with CF often have lung infections that occur repeatedly or worsen over time. The lung infections are often caused by PA. Treatment with antibiotics is used to reduce the presence of the bacteria. The antibiotics may be given orally, intravenously, or inhaled as a mist. The purpose of this study was to evaluate whether AZLI, an investigational formulation of the antibiotic aztreonam, is safe in repeated courses in patients with CF and PA.

A course of AZLI treatment in this study comprised 28 days, followed by a 28-day period off treatment. Participants could receive up to 9 courses of AZLI, with a total time on study of up to 18 months. Safety and efficacy results for the 18-month, 9-course period are reported, with efficacy results presented on a by-treatment course basis.

ELIGIBILITY:
Inclusion Criteria:

* Compliance with Studies CP-AI-005 (NCT00104520) or CP-AI-007 (NCT00112359) by taking at least 50% of expected study medication.
* Completion of CP-AI-005 or CP-AI-007 or was withdrawn due to need for antipseudomonal antibiotics or for an AE unrelated to study medication tolerance.
* Ability to provide written informed consent/assent prior to initiation of study-related procedures.
* Ability to perform reproducible pulmonary function tests.

Exclusion Criteria:

* Use of any investigational medication or device between the last visit of CP-AI-005 or CP-AI-007 and Visit 1 of this study.
* Concurrent participation in a study of another investigational drug or device.
* Current use of oral corticosteroids in doses exceeding the equivalent of 10 mg prednisone/day or 20 mg prednisone every other day.
* History of sputum or throat swab culture yielding Burkholderia cepacia in the previous 2 years.
* History of daily continuous oxygen supplementation or requirement for more than 2 liters/minute at night.
* Inability to tolerate study medication in CP-AI-005 or CP-AI-007.
* Known local or systemic hypersensitivity to aztreonam.
* Inability to tolerate inhalation of a short acting beta-2 agonist.
* Abnormal renal or hepatic function based on results of most recent test.
* Female of child-bearing potential who was pregnant, lactating, or not (in the opinion of the investigator) practicing an acceptable method of birth control.
* Any serious or active medical or psychiatric illness which, in the opinion of the investigator, would have interfered with participant treatment, assessment, or compliance with the protocol.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2005-08; Primary Completion 2008-11 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Montgomery, MD, Study Director — Gilead Sciences
Locations (65):
- United States (56):
  - Birmingham, Alabama
  - Anchorage, Alaska
  - Phoenix, Arizona
  - Little Rock, Arkansas
  - La Jolla, California
  - Los Angeles, California
  - Oakland, California
  - Orange, California
  - Denver, Colorado
  - Hartford, Connecticut
  - New Haven, Connecticut
  - Jacksonville, Florida
  - Orlando, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Chicago, Illinois
  - Glenview, Illinois
  - Maywood, Illinois
  - Park Ridge, Illinois
  - Indianapolis, Indiana
  - Wichita, Kansas
  - Shreveport, Louisiana
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Detroit, Michigan
  - Minneapolis, Minnesota
  - Columbia, Missouri
  - St Louis, Missouri
  - Las Vegas, Nevada
  - Livingston, New Jersey
  - Morristown, New Jersey
  - Albany, New York
  - Brooklyn, New York
  - Buffalo, New York
  - New Hyde Park, New York
  - New York, New York
  - Syracuse, New York
  - Valhalla, New York
  - Chapel Hill, North Carolina
  - Akron, Ohio
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Dayton, Ohio
  - Oklahoma City, Oklahoma
  - Hershey, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Charleston, South Carolina
  - Columbia, South Carolina
  - Houston, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Portsmouth, Virginia
  - Richmond, Virginia
  - Seattle, Washington
  - Morgantown, West Virginia
- Australia (6):
  - Westmead, New South Wales
  - Herston, Queensland
  - Adelaide, South Australia
  - Prahan, Victoria
  - Nedlands, Western Australia
  - Perth, Western Australia
- Canada (2):
  - Edmonton, Alberta
  - London, Ontario
- Auckland, New Zealand

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Open-label, Phase 3 follow-on study for participants from Studies CP-AI-005 (NCT00104520) and CP-AI-007 (NCT00112359). Participants were enrolled at 71 sites in the United States, Canada, Australia, and New Zealand. The date of first enrollment was 17 August 2005, and the date of database lock was 23 January 2009.
Pre-assignment Details: Participants enrolled in this study were required to have previously participated in CP-AI-005 or CP-AI-007. Participants from CP-AI-005 received open-label AZLI (75 mg) in the same regimen (twice daily [BID] or three times daily [TID]) to which they were previously randomized. Participants from CP-AI-007 received open-label AZLI (75 mg) TID.
Groups:
- 75 mg AZLI Two Times a Day (BID): Participants received up to 9 treatment courses of open-label 75 mg AZLI BID via an investigational nebulizer; each treatment course consisted of 28 days of AZLI and was followed by a 28-day interval off therapy.
  BID = twice daily
- 75 mg AZLI Three Times a Day (TID): Participants received up to 9 treatment courses of open-label 75 mg AZLI TID via an investigational nebulizer; each treatment course consisted of 28 days of AZLI and was followed by a 28-day interval off therapy.
  TID = three times daily
Period: Overall Study
Arm/Group | 75 mg AZLI Two Times a Day (BID) | 75 mg AZLI Three Times a Day (TID)
Started | 85 | 189
Completed | 65 | 130
Not Completed | 20 | 59
Not completed — AE unrelated to study | 2 | 9
Not completed — Study drug intolerance (AE) | 2 | 8
Not completed — AE related to study | 1 | 4
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 1 | 5
Not completed — Noncompliance | 0 | 5
Not completed — Personal or administrative | 10 | 22
Not completed — Withdrawal by Subject | 3 | 5
Not completed — Pregnancy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 75 mg AZLI Two Times a Day (BID) | 75 mg AZLI Three Times a Day (TID) | Total
Number analyzed (Participants) | 85 | 189 | 274
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 19 | 36 | 55
  Between 18 and 65 years | 65 | 151 | 216
  >=65 years | 1 | 2 | 3
Age Continuous [Mean (Standard Deviation); unit: years] | 27.3 (11.4) | 29.0 (13.0) | 28.5 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 89 | 123
  Male | 51 | 100 | 151
Region of Enrollment [Number; unit: participants]
  United States | 85 | 157 | 242
  Canada | 0 | 8 | 8
  Australia | 0 | 22 | 22
  New Zealand | 0 | 2 | 2
Aztreonam Minimum Inhibitory Concentration (MIC) for Pseudomonas aeruginosa (PA) [Number; unit: participants] — Number of partipipants with an MIC of aztreonam ≤ 8 µg/mL or >8 µg/mL for PA are summarized.
  participants
    Aztreonam MIC > 8 µg/mL | 30 | 72 | 102
    Aztreonam MIC < or = 8 µg/mL | 46 | 99 | 145
    Unknown | 9 | 18 | 27
Disease severity as defined by FEV1 percent predicted category [Number; unit: Participants] — FEV1 percent predicted is a normalized value of FEV1 calculated using the Knudson equation and based upon participant age, gender, and height. This baseline measure indicates the number of subjects with FEV1 greater than 50% and less than or equal to 50% of the predicted value based on age, gender, and height at screening.
  Participants
    FEV1 > 50% predicted | 49 | 114 | 163
    FEV1 ≤ 50% predicted | 36 | 74 | 110
    Unknown | 0 | 1 | 1
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 21.30 (3.25) | 21.44 (3.96) | 21.40 (3.75)
Cystic Fibrosis Questionnaire-Revised Respiratory Symptom Score (CFQ-R RSS) [Mean (Standard Deviation); unit: Units on a scale] — CFQ-R RSS scale range 0-100, with higher scores indicating fewer CF symptoms.
  Units on a scale | 65.410 (16.896) | 60.332 (18.497) | 61.895 (18.141)
Forced Expiratory Volume in 1 Second (FEV1) Percent Predicted [Mean (Standard Deviation); unit: Percent] — FEV1 percent predicted is a normalized value of FEV1 calculated using the Knudson equation and based upon participant age, gender, and height.
  Percent | 56.711 (17.505) | 55.071 (15.428) | 55.582 (16.089)
Log10 Pseudomonas aeruginosa (PA) Colony-Forming Units (CFUs) in Sputum [Mean (Standard Deviation); unit: log10 CFUs/g] | 5.71 (2.249) | 6.16 (1.894) | 6.02 (2.014)
Weight [Mean (Standard Deviation); unit: kg] | 59.52 (13.28) | 59.28 (15.81) | 59.36 (15.05)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Adverse Events (AEs)
Description: Participants experiencing at least 1 treatment-emergent AE or at least 1 serious adverse event (SAE) were summarized for the study as a whole. A treatment-emergent AE was any physical or clinical worsening in symptoms or disease experienced by the participant, whether or not the event was considered related to study participation or study procedures. An SAE was any adverse experience that resulted in hospitalization or death.
  Participants were monitored for AEs and SAEs during all on-treatment and off-treatment intervals throughout the 18-month study period.
Time Frame: Overall study (72 weeks) included nine 28-day courses of study drug alternating with nine 28-day courses off drug
Population: The analysis population consisted of all enrolled participants who received one or more doses of AZLI.
Measure: Number; unit: participants
Arm/Group | 75 mg AZLI Two Times a Day (BID) | 75 mg AZLI Three Times a Day (TID)
Number analyzed (Participants) | 85 | 189
participants
  Number of Participants Reporting at Least One AE | 83 | 185
  Participants Reporting at least One Related AE | 30 | 79
  Number of Participants Reporting at Least One SAE | 38 | 100
  Participants with Study Drug Withdrawn due to AE | 7 | 38
  Number of Participants who Died on Study | 1 | 0

2. Primary Outcome: Number of Subjects With <15% or ≥15% Decline in Forced Expiratory Volume in 1 Second [FEV1] From Pretreatment to 30 Minutes After Treatment With AZLI
Description: Airway reactivity (percent change in FEV1 from pretreatment to 30 minutes after treatment with AZLI) was assessed at all study visits in which a participant received AZLI treatment. A participant was included in this endpoint if they experienced a decline in FEV1 of ≥15% at any visit in which they received AZLI.
Time Frame: Overall study (72 weeks) included nine 28-day courses of study drug alternating with nine 28-day courses off drug
Population: The analysis population consisted of all enrolled participants who received one or more doses of AZLI.
Measure: Number; unit: Participants
Arm/Group | 75 mg AZLI Two Times a Day (BID) | 75 mg AZLI Three Times a Day (TID)
Number analyzed (Participants) | 85 | 189
Participants
  Participants with <15% decline | 76 | 175
  Participants with >=15% decline | 9 | 14

3. Primary Outcome: Change in Heart Rate (HR)
Description: HR was recorded at all visits.
  Change from baseline at the end of AZLI treatment Courses 1 (Visit 2), 3 (Visit 4), and 9 (Visit 19) was determined.
Time Frame: Baseline, and end of treatment Courses 1 (Week 4), 3 (Week 20) and 9 (Week 68)
Population: The analysis population consisted of all enrolled participants who received one or more doses of AZLI.
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | 75 mg AZLI Two Times a Day (BID) | 75 mg AZLI Three Times a Day (TID)
Number analyzed (Participants) | 85 | 189
beats/minute
  HR, End of Treatment Course 1 | 1.08 (15.9) | -0.07 (12.9)
  HR, End of Treatment Course 3 | -0.53 (13.7) | 0.13 (14.5)
  HR, End of Treatment Course 9 | 3.87 (12.9) | -0.06 (12.5)

4. Primary Outcome: Change in Systolic and Diastolic Blood Pressure (BP)
Description: BP was recorded at all visits.
  Change from baseline at the end of AZLI treatment Courses 1 (Visit 2), 3 (Visit 4), and 9 (Visit 19) was determined.
Time Frame: Baseline, and end of treatment Courses 1 (Week 4), 3 (Week 20) and 9 (Week 68)
Population: The analysis population consisted of all enrolled participants who received one or more doses of AZLI.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | 75 mg AZLI Two Times a Day (BID) | 75 mg AZLI Three Times a Day (TID)
Number analyzed (Participants) | 85 | 189
mm Hg
  Systolic BP, End of Treatment Course 1 | 0.75 (11.0) | 1.19 (11.7)
  Systolic BP, End of Treatment Course 3 | -0.67 (13.1) | 0.29 (11.9)
  Systolic BP, End of Treatment Course 9 | -1.06 (13.2) | -0.33 (11.0)
  Diastolic BP, End of Treatment Course 1 | 0.49 (8.4) | 0.05 (8.2)
  Diastolic BP, End of Treatment Course 3 | -1.64 (8.7) | -0.89 (8.3)
  Diastolic BP, End of Treatment Course 9 | -0.40 (9.4) | -0.76 (10.0)

5. Secondary Outcome: Change From Baseline in Pseudomonas Aeruginosa (PA) log10 Colony-forming Units (CFU) Per Gram of Sputum
Description: Sputum samples were collected at all participant visits of the study for analysis of microbiology endpoints. Sputum samples were processed for qualitative and quantitative culture of PA (each morphotype).
  Due to the skewness of the distribution of CFU data, the data were transformed using the base 10 logarithm, in an attempt to normalize the data and allow for parametric tests, before calculating changes. To account for zero values, 1 was added to each CFU measurement before being transformed. Any CFU data values where PA was not isolated from a valid culture were set to zero.
Time Frame: Baseline, and the end of treatment Courses 1 (Week 4), 3 (Week 20), and 9 (Week 68)
Population: The analysis population consisted of all enrolled participants who received one or more doses of AZLI.
Measure: Mean (Standard Deviation); unit: Log10 PA CFUs/g
Arm/Group | 75 mg AZLI Two Times a Day (BID) | 75 mg AZLI Three Times a Day (TID)
Number analyzed (Participants) | 85 | 189
Log10 PA CFUs/g
  End of Treatment Course 1 | -0.20 (1.5) | -0.81 (1.8)
  End of Treatment Course 3 | -0.43 (1.4) | -0.53 (2.1)
  End of Treatment Course 9 | -0.47 (1.9) | -0.60 (2.1)

6. Secondary Outcome: Number of Participants With Other Pathogens
Description: Sputum samples were collected at all study visits for qualitative and quantitative culture for Burkholderia cepacia complex (BCC), Stenotrophomonas maltophilia, Achromobacter xylosoxidans, Staphylococcus aureus (including methicillin-sensitive [MSSA] and methicillin-resistant [MRSA] S.aureus), and fungal organisms.
  Number of participants with other pathogens at baseline and end of AZLI treatment Courses 1, 3, and 9 are reported.
Time Frame: Baseline; end of treatment Courses 1 (Week 4), 3 (Week 20), and 9 (Week 68); and at Follow-up (Week 72)
Population: The analysis population consisted of all enrolled participants who received one or more doses of AZLI.
Measure: Number; unit: Participants
Arm/Group | 75 mg AZLI Two Times a Day (BID) | 75 mg AZLI Three Times a Day (TID)
Number analyzed (Participants) | 85 | 189
Participants
  S. aureus, Baseline | 33 | 65
  S. aureus, End of Treatment Course 1 | 34 | 66
  S. aureus, End of Treatment Course 3 | 41 | 68
  S. aureus, End of Treatment Course 9 | 15 | 51
  S. aureus, Follow-up | 16 | 49
  MSSA, Baseline | 26 | 32
  MSSA, End of Treatment Course 1 | 27 | 32
  MSSA, End of Treatment Course 3 | 31 | 35
  MSSA, End of Treatment Course 9 | 10 | 31
  MSSA, Follow-up | 11 | 32
  MRSA, Baseline | 7 | 25
  MRSA, End of Treatment Course 1 | 7 | 25
  MRSA, End of Treatment Course 3 | 9 | 26
  MRSA, End of Treatment Course 9 | 5 | 19
  MRSA, Follow-up | 5 | 17
  BCC, Baseline | 0 | 1
  BCC, End of Treatment Course 1 | 0 | 0
  BCC, End of Treatment Course 3 | 0 | 1
  BCC, End of Treatment Course 9 | 0 | 0
  BCC, Follow-up | 0 | 1
  S. maltophilia, Baseline | 13 | 14
  S. maltophilia, End of Treatment Course 1 | 12 | 17
  S. maltophilia, End of Treatment Course 3 | 11 | 15
  S. maltophilia, End of Treatment Course 9 | 5 | 14
  S. maltophilia, Follow-up | 6 | 12
  A. xylosoxidans, Baseline | 8 | 13
  A. xylosoxidans, End of Treatment Course 1 | 8 | 11
  A. xylosoxidans, End of Treatment Course 3 | 7 | 12
  A. xylosoxidans, End of Treatment Course 9 | 4 | 9
  A. xylosoxidans, Follow-up | 4 | 7
  Aspergillus Species, Baseline | 15 | 41
  Aspergillus Species, End of Treatment Course 1 | 18 | 35
  Aspergillus Species, End of Treatment Course 3 | 21 | 33
  Aspergillus Species, End of Treatment Course 9 | 9 | 27
  Aspergillus Species, Follow-up | 10 | 38
  Candida Species, Baseline | 51 | 135
  Candida Species, End of Treatment Course 1 | 48 | 139
  Candida Species, End of Treatment Course 3 | 55 | 125
  Candida Species, End of Treatment Course 9 | 38 | 101
  Candida Species, Follow-up | 36 | 95

7. Secondary Outcome: Minimum Inhibitory Concentration (MIC) of Aztreonam
Description: The aztreonam susceptibility of PA isolates from expectorated sputum samples (collected at all visits) was assessed.
  MIC50 = minimum inhibitory concentration (minimum concentration of an agent that inhibits 50% of isolates from a particular organism).
  MIC90 = minimum inhibitory concentration (minimum concentration of an agent that inhibits 90% of isolates from a particular organism).
  MIC50 and MIC90 values are single measurements for the entire population and not measured on a per-participant basis.
Time Frame: Baseline; end of treatment Courses 1 (Week 4), 3 (Week 20), and 9 (Week 68); and at Follow-up (Week 72)
Population: The analysis population consisted of all enrolled participants who received one or more doses of AZLI.
Measure: Number; unit: µg/mL
Arm/Group | 75 mg AZLI Two Times a Day (BID) | 75 mg AZLI Three Times a Day (TID)
Number analyzed (Participants) | 85 | 189
µg/mL
  MIC50, Baseline | 4 | 4
  MIC50, End of Treatment Course 1 | 4 | 8
  MIC50, End of Treatment Course 3 | 8 | 8
  MIC50, End of Treatment Course 9 | 16 | 8
  MIC50, Follow-up | 4 | 8
  MIC90, Baseline | 128 | 128
  MIC90, End of Treatment Course 1 | 256 | 256
  MIC90, End of Treatment Course 3 | 256 | 256
  MIC90, End of Treatment Course 9 | 512 | 512
  MIC90, Follow-up | 128 | 256

8. Secondary Outcome: Percent Change in Pulmonary Function (FEV1, FEV1 Percent Predicted, FVC, FEF25-75)
Description: Spirometry was performed at each visit. FEV1, FVC, and FEF25-75 were recorded at all visits according to American Thoracic Society (ATS) guidelines.
  FEV1 = the volume of air exhaled in 1 second. FEV1 % predicted is a normalized value of FEV1 calculated using the Knudson equation, based upon participant age, gender, and height. FVC = (forced vital capacity) the maximal volume of air exhaled with maximally forced effort from a position of maximal inspiration. FEF25-75 = forced expiratory flow from 25% to 75% of the FVC.
  The percent change from baseline is presented for each endpoint.
Time Frame: Baseline, and end of treatment Courses 1 (Week 4), 3 (Week 20), and 9 (Week 68)
Population: The analysis population consisted of all enrolled participants who received one or more doses of AZLI.
Measure: Mean (Standard Deviation); unit: Percent change from baseline
Arm/Group | 75 mg AZLI Two Times a Day (BID) | 75 mg AZLI Three Times a Day (TID)
Number analyzed (Participants) | 85 | 189
Percent change from baseline
  FEV1 (L), End of Treatment Course 1 | 4.87 (11.428) | 7.98 (16.512)
  FEV1 (L), End of Treatment Course 3 | 3.55 (12.491) | 6.04 (16.489)
  FEV1 (L), End of Treatment Course 9 | 1.31 (15.924) | 3.98 (17.899)
  FEV1 Percent Predicted, End of Treatment Course 1 | 4.91 (11.599) | 7.97 (16.511)
  FEV1 Percent Predicted, End of Treatment Course 3 | 3.46 (12.504) | 6.15 (16.592)
  FEV1 Percent Predicted, End of Treatment Course 9 | 1.23 (15.673) | 4.24 (17.992)
  FVC (L), End of Treatment Course 1 | 3.13 (11.946) | 5.59 (16.533)
  FVC (L), End of Treatment Course 3 | 1.77 (10.948) | 5.95 (13.178)
  FVC (L), End of Treatment Course 9 | 1.51 (14.150) | 5.29 (14.075)
  FEF25-75 (L/sec), End of Treatment Course 1 | 12.81 (36.149) | 14.14 (36.089)
  FEF25-75 (L/sec), End of Treatment Course 3 | 16.05 (55.447) | 4.81 (32.579)
  FEF25-75 (L/sec), End of Treatment Course 9 | 3.24 (28.506) | 3.29 (36.329)

9. Secondary Outcome: Change in Clinical Symptoms as Assessed by the Cystic Fibrosis Questionnaire-Revised Respiratory Symptom Scale (CFQ-R RSS)
Description: The CFQ-R was administered at baseline and every visit thereafter. The endpoint was change in respiratory symptoms from baseline, assessed with the CFQ-R RSS (range of scores: 0-100; higher scores indicate fewer symptoms). The minimal clinically important difference (MCID) corresponds to the smallest change in symptoms that a patient can detect and is a change in score of 4 points.
Time Frame: Baseline, and end of treatment Courses 1 (Week 4), 3 (Week 20), and 9 (Week 68)
Population: The analysis population consisted of all enrolled participants who received one or more doses of AZLI.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | 75 mg AZLI Two Times a Day (BID) | 75 mg AZLI Three Times a Day (TID)
Number analyzed (Participants) | 85 | 189
Units on a scale
  End of Treatment Course 1 | 3.53 (12.243) | 6.83 (17.379)
  End of Treatment Course 3 | 0.37 (19.296) | 7.34 (18.518)
  End of Treatment Course 9 | 0.30 (15.217) | 6.01 (17.943)

10. Secondary Outcome: Time to First Hospitalization Due to a Respiratory Event
Description: Details of all hospitalizations, including the dates of admission and discharge, were recorded on the serious adverse event (SAE) electronic case report form (eCRF).
  Time to first hospitalization was the number of days from baseline (Visit 1) to the date of first hospitalization or the date of study completion (last visit) /or early withdrawal if censored.
Time Frame: Overall study (72 weeks) included nine 28-day courses of study drug alternating with nine 28-day courses off drug
Population: The analysis population consisted of all enrolled participants who received one or more doses of AZLI.
Measure: Median (Full Range); unit: Days
Arm/Group | 75 mg AZLI Two Times a Day (BID) | 75 mg AZLI Three Times a Day (TID)
Number analyzed (Participants) | 85 | 189
Days | 359 (27.60) [4 to 431] | 417 (21.32) [1 to 609]

11. Secondary Outcome: Change in Body Weight
Description: Weight was measured at all visits and was reported to the nearest 0.1 kg/lb. Percent change in weight from baseline was calculated.
Time Frame: Baseline, and end of treatment Courses 1 (Week 4), 3 (Week 20), and 9 (Week 68)
Population: The analysis population consisted of all enrolled participants who received one or more doses of AZLI.
Measure: Mean (Standard Error); unit: Percent change from baseline
Arm/Group | 75 mg AZLI Two Times a Day (BID) | 75 mg AZLI Three Times a Day (TID)
Number analyzed (Participants) | 85 | 189
Percent change from baseline
  End of Treatment Course 1 | 0.58 (2.449) | 0.85 (2.338)
  End of Treatment Course 3 | 1.31 (3.769) | 1.38 (3.991)
  End of Treatment Course 9 | 3.24 (6.542) | 3.55 (7.431)

12. Secondary Outcome: Missed School/Work Days Due to CF Symptoms
Description: Participants were provided with a diary card at each visit to record days of work and/or school missed due to their CF symptoms.
  The percentage of school/work days missed was calculated as the total number of school/work days missed divided by the total number of on-study days multiplied by 100 across all participants in a treatment group.
Time Frame: Overall study (72 weeks) included nine 28-day courses of study drug alternating with nine 28-day courses off drug
Population: The analysis population consisted of all enrolled participants who received one or more doses of AZLI.
Measure: Mean (Standard Deviation); unit: Percentage of days missed
Arm/Group | 75 mg AZLI Two Times a Day (BID) | 75 mg AZLI Three Times a Day (TID)
Number analyzed (Participants) | 85 | 189
Percentage of days missed | 2.00 (4.04) | 3.19 (6.86)

13. Secondary Outcome: Time to Intravenous (IV) Antipseudomonal Antibiotics
Description: Use of IV antipseudomonal antibiotics was compiled from data recorded on the Concomitant Medications eCRF. The time to first IV antipseudomonal antibiotic use was the number of days from baseline (Visit 1) to the date of first IV antipseudomonal antibiotic use or the date of study completion (last visit) /or early withdrawal if censored.
Time Frame: Overall study (72 weeks) included nine 28-day courses of study drug alternating with nine 28-day courses off drug
Population: The analysis population consisted of all enrolled participants who received one or more doses of AZLI.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | 75 mg AZLI Two Times a Day (BID) | 75 mg AZLI Three Times a Day (TID)
Number analyzed (Participants) | 85 | 189
Days | 276 [217 to 316] | 232 [179 to 288]

14. Primary Outcome: Change in Temperature
Description: Temperature was recorded at all visits.
  Change from baseline at the end of AZLI treatment Courses 1 (Visit 2), 3 (Visit 4), and 9 (Visit 19) was determined.
Time Frame: Baseline, and end of treatment Courses 1 (Week 4), 3 (Week 20) and 9 (Week 68)
Population: The analysis population consisted of all enrolled participants who received one or more doses of AZLI.
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | 75 mg AZLI Two Times a Day (BID) | 75 mg AZLI Three Times a Day (TID)
Number analyzed (Participants) | 85 | 189
degrees Celsius
  Temperature (Celsius) End of Treatment Course 1 | -0.05 (0.4) | 0.00 (0.5)
  Temperature (Celsius) End of Treatment Course 3 | -0.09 (0.4) | 0.01 (0.5)
  Temperature (Celsius) End of Treatment Course 9 | 0.04 (0.6) | 0.05 (0.5)

15. Primary Outcome: Change in Respiratory Rate (RR)
Description: RR was recorded at all visits.
  Change from baseline at the end of AZLI treatment Courses 1 (Visit 2), 3 (Visit 4), and 9 (Visit 19) was determined.
Time Frame: Baseline, and end of treatment Courses 1 (Week 4), 3 (Week 20) and 9 (Week 68)
Population: The analysis population consisted of all enrolled participants who received one or more doses of AZLI.
Measure: Mean (Standard Deviation); unit: breaths/minute
Arm/Group | 75 mg AZLI Two Times a Day (BID) | 75 mg AZLI Three Times a Day (TID)
Number analyzed (Participants) | 85 | 189
breaths/minute
  RR, End of Treatment Course 1 | -0.07 (2.8) | 0.17 (3.9)
  RR, End of Treatment Course 3 | -0.03 (3.3) | 0.02 (3.7)
  RR, End of Treatment Course 9 | 0.02 (3.8) | 0.33 (3.3)

16. Primary Outcome: Serum Hematology - Concentration of White Blood Cells (WBC), Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, and Platelets
Time Frame: Baseline and end of Course 9 (Week 68)
Population: The analysis population consisted of all enrolled participants who received one or more doses of AZLI. Results obtained at the end of a 28-day treatment period are presented for selected timepoints.
Measure: Mean (Standard Deviation); unit: number of cells x10^3/µL
Arm/Group | 75 mg AZLI Two Times a Day (BID) | 75 mg AZLI Three Times a Day (TID)
Number analyzed (Participants) | 85 | 189
number of cells x10^3/µL
  WBCs, Baseline | 9.28 (3.692) | 10.11 (3.635)
  WBCs, End of Treatment Course 9 | 9.47 (3.998) | 9.53 (3.562)
  Basophils, Baseline | 0.05 (0.037) | 0.06 (0.144)
  Basophils, End of Treatment Course 9 | 0.05 (0.034) | 0.05 (0.033)
  Eosinophils, Baseline | 0.18 (0.111) | 0.19 (0.152)
  Eosinophils, End of Treatment Course 9 | 0.21 (0.209) | 0.17 (0.144)
  Lymphocytes, Baseline | 2.00 (0.623) | 2.17 (0.732)
  Lymphocytes, End of Treatment Course 9 | 1.99 (0.801) | 2.13 (0.719)
  Monocytes, Baseline | 0.47 (0.190) | 0.54 (0.241)
  Monocytes, End of Treatment Course 9 | 0.50 (0.157) | 0.52 (0.210)
  Neutrophils, Baseline | 6.54 (3.295) | 7.09 (3.227)
  Neutrophils, End of Treatment Course 9 | 6.68 (3.481) | 6.63 (3.345)
  Platelets, Baseline | 293.11 (85.681) | 340.19 (106.749)
  Platelets, End of Treatment Course 9 | 290.43 (106.903) | 311.39 (98.370)

17. Primary Outcome: Serum Hematology - Percent of Differential for Basophils, Eosinophils, Lymphocytes, Monocytes, and Neutrophils
Time Frame: Baseline and end of treatment Course 9 (Week 68)
Population: The analysis population consisted of all enrolled participants who received one or more doses of AZLI.
Measure: Mean (Standard Deviation); unit: percent of differential
Arm/Group | 75 mg AZLI Two Times a Day (BID) | 75 mg AZLI Three Times a Day (TID)
Number analyzed (Participants) | 85 | 189
percent of differential
  Basophils, Baseline | 0.59 (0.379) | 0.61 (0.390)
  Basophils, End of Treatment Course 9 | 0.59 (0.393) | 0.62 (0.340)
  Eosinophils, Baseline | 2.05 (1.194) | 1.95 (1.453)
  Eosinophils, End of Treatment Course 9 | 2.20 (1.694) | 1.88 (1.625)
  Lymphocytes, Baseline | 23.40 (8.278) | 22.74 (8.265)
  Lymphocytes, End of Treatment Course 9 | 22.30 (7.462) | 24.17 (8.441)
  Monocytes, Baseline | 5.32 (1.919) | 5.26 (1.752)
  Monocytes, End of Treatment Course 9 | 5.64 (1.660) | 5.77 (1.977)
  Neutrophils, Baseline | 68.39 (9.331) | 69.26 (9.261)
  Neutrophils, End of Treatment Course 9 | 69.02 (8.551) | 67.46 (9.808)

18. Primary Outcome: Serum Hematology - Number of Red Blood Cells (RBC)
Time Frame: Baseline and end of treatment Course 9 (Week 68)
Population: The analysis population consisted of all enrolled participants who received one or more doses of AZLI.
Measure: Mean (Standard Deviation); unit: number x10^6/µL
Arm/Group | 75 mg AZLI Two Times a Day (BID) | 75 mg AZLI Three Times a Day (TID)
Number analyzed (Participants) | 85 | 189
number x10^6/µL
  RBCs, Baseline | 5.15 (0.442) | 4.94 (0.499)
  RBCs, End of treatment 9 | 4.93 (0.376) | 4.77 (0.492)

19. Primary Outcome: Serum Hematology - Hematocrit
Time Frame: Baseline and end of treatment Course 9 (Week 68)
Population: The analysis population consisted of all enrolled participants who received one or more doses of AZLI.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | 75 mg AZLI Two Times a Day (BID) | 75 mg AZLI Three Times a Day (TID)
Number analyzed (Participants) | 85 | 189
percent
  Hematocrit, Baseline | 43.43 (4.037) | 42.45 (4.142)
  Hematocrit, End of treatment course 9 | 42.00 (3.317) | 41.63 (4.056)

20. Primary Outcome: Serum Hematology - Hemoglobin
Time Frame: Baseline and end of treatment Course 9 (Week 68)
Population: The analysis population consisted of all enrolled participants who received one or more doses of AZLI.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | 75 mg AZLI Two Times a Day (BID) | 75 mg AZLI Three Times a Day (TID)
Number analyzed (Participants) | 85 | 189
g/dL
  Hemoglobin, Baseline | 14.06 (1.406) | 13.70 (1.448)
  Hemoglobin, End of treatment course 9 | 13.89 (1.195) | 13.71 (1.475)

21. Primary Outcome: Serum Hematology - Mean Corpuscular Volume (MCV)
Time Frame: Baseline and end of treatment Course 9 (Week 68)
Population: The analysis population consisted of all enrolled participants who received one or more doses of AZLI.
Measure: Mean (Standard Deviation); unit: fL
Arm/Group | 75 mg AZLI Two Times a Day (BID) | 75 mg AZLI Three Times a Day (TID)
Number analyzed (Participants) | 85 | 189
fL
  MCV, Baseline | 84.33 (4.880) | 86.08 (5.560)
  MCV, End of treatment course 9 | 85.38 (5.232) | 87.72 (5.450)

22. Primary Outcome: Serum Hematology - Mean Corpuscular Hemoglobin (MCH)
Time Frame: Baseline and end of treatment Course 9 (Week 68)
Population: The analysis population consisted of all enrolled participants who received one or more doses of AZLI.
Measure: Mean (Standard Deviation); unit: pg
Arm/Group | 75 mg AZLI Two Times a Day (BID) | 75 mg AZLI Three Times a Day (TID)
Number analyzed (Participants) | 85 | 189
pg
  MCH, Baseline | 27.43 (1.824) | 27.84 (2.090)
  MCH, End of treatment course 9 | 28.35 (2.282) | 28.89 (2.050)

23. Primary Outcome: Serum Hematology - Mean Corpuscular Hemoglobin Concentration (MCHC)
Time Frame: Baseline and end of treatment Course 9 (Week 68)
Population: The analysis population consisted of all enrolled participants who received one or more doses of AZLI.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | 75 mg AZLI Two Times a Day (BID) | 75 mg AZLI Three Times a Day (TID)
Number analyzed (Participants) | 85 | 189
g/dL
  MCHC, Baseline | 32.41 (1.032) | 32.34 (1.228)
  MCHC, End of treatment course 9 | 33.13 (1.272) | 32.99 (1.288)

24. Primary Outcome: Serum Chemistry - Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), and Gamma-glutamlytransferase (GGT)
Time Frame: Baseline and end of treatment Course 9 (Week 68)
Population: The analysis population consisted of all enrolled participants who received one or more doses of AZLI.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | 75 mg AZLI Two Times a Day (BID) | 75 mg AZLI Three Times a Day (TID)
Number analyzed (Participants) | 85 | 189
U/L
  ALT, Baseline | 31.21 (22.343) | 26.65 (18.982)
  ALT, End of Treatment Course 9 | 30.78 (24.045) | 27.81 (21.794)
  AST, Baseline | 27.83 (14.856) | 25.77 (15.556)
  AST, End of Treatment Course 9 | 26.84 (14.588) | 26.22 (15.240)
  GGT, Baseline | 35.49 (48.215) | 29.64 (41.862)
  GGT, End of Treatment Course 9 | 40.83 (57.471) | 32.39 (39.662)

25. Primary Outcome: Serum Chemistry - Concentration of Calcium, Creatinine, Direct Bilirubin, Total Bilirubin, Serum Glucose, and Blood Urea Nitrogen
Time Frame: Baseline and end of treatment Course 9 (Week 68)
Population: The analysis population consisted of all enrolled participants who received one or more doses of AZLI.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | 75 mg AZLI Two Times a Day (BID) | 75 mg AZLI Three Times a Day (TID)
Number analyzed (Participants) | 85 | 189
mg/dL
  Calcium (EDTA), Baseline | 9.67 (0.406) | 9.56 (0.416)
  Calcium (EDTA), End of Treatment Course 9 | 9.43 (0.385) | 9.47 (0.427)
  Creatinine, Baseline | 0.80 (0.202) | 0.81 (0.317)
  Creatinine, End of Treatment Course 9 | 0.80 (0.207) | 0.82 (0.295)
  Direct bilirubin, Baseline | 0.14 (0.076) | 0.13 (0.064)
  Direct bilirubin, End of Treatment Course 9 | 0.16 (0.081) | 0.14 (0.072)
  Total bilirubin, Baseline | 0.42 (0.237) | 0.43 (0.298)
  Total bilirubin, End of Treatment Course 9 | 0.51 (0.294) | 0.49 (0.377)
  Serum glucose, Baseline | 115.46 (55.211) | 111.53 (49.485)
  Serum glucose, End of Treatment Course 9 | 121.11 (57.47) | 116.40 (65.046)
  BUN, Baseline | 14.65 (4.258) | 14.32 (5.698)
  BUN, End of Treatment Course 9 | 13.83 (4.764) | 14.49 (4.805)

26. Primary Outcome: Serum Chemistry - Concentration of Chloride, Potassium, and Sodium
Time Frame: Baseline and end of treatment Course 9 (Week 68)
Population: The analysis population consisted of all enrolled participants who received one or more doses of AZLI.
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | 75 mg AZLI Two Times a Day (BID) | 75 mg AZLI Three Times a Day (TID)
Number analyzed (Participants) | 85 | 189
mEq/L
  Serum chloride, Baseline | 102.17 (2.904) | 102.22 (2.943)
  Serum chloride, End of Treatment Course 9 | 101.81 (2.610) | 102.16 (2.977)
  Serum potassium, Baseline | 4.20 (0.354) | 4.29 (0.370)
  Serum potassium, End of Treatment Course 9 | 4.19 (0.388) | 4.25 (0.372)
  Serum sodium, Baseline | 139.18 (2.984) | 139.23 (2.618)
  Serum sodium, End of Treatment Course 9 | 138.64 (2.608) | 138.88 (2.694)

27. Primary Outcome: Serum Chemistry - Concentration of Total Protein
Time Frame: Baseline and end of treatment Course 9 (Week 68)
Population: The analysis population consisted of all enrolled participants who received one or more doses of AZLI.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | 75 mg AZLI Two Times a Day (BID) | 75 mg AZLI Three Times a Day (TID)
Number analyzed (Participants) | 85 | 189
g/dL
  Total protein, Baseline | 7.63 (0.588) | 7.58 (0.536)
  Total protein, End of Treatment Course 9 | 7.47 (0.425) | 7.53 (0.560)

ADVERSE EVENTS:
Time Frame: Participants were monitored for AEs and SAEs during all on-treatment and off-treatment intervals. Participants could receive up to 9 courses of AZLI, with total time on study of up to 18 months. Events occurring during the 18-month period are reported.
Description: A treatment-emergent AE was any physical or clinical worsening in symptoms or disease experienced by the participant at any time during the course of the study, whether or not the event was considered related to study participation or study procedures. An SAE was any adverse experience that resulted in death or hospitalization.
Arm/Group | 75 mg AZLI Two Times a Day (BID) | 75 mg AZLI Three Times a Day (TID)
Serious Adverse Events (participants affected / at risk) | 38/85 | 100/189
Other Adverse Events (participants affected / at risk) | 83/85 | 185/189
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 75 mg AZLI Two Times a Day (BID) (N=85) | 75 mg AZLI Three Times a Day (TID) (N=189)
Abdominal pain (Gastrointestinal disorders) | 4 | 7
Abdominal pain lower (Gastrointestinal disorders) | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 5
Abdominal tenderness (Gastrointestinal disorders) | 0 | 2
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 4
Antibacterial prophylaxis (Surgical and medical procedures) | 2 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Asthenia (General disorders) | 1 | 4
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Blood chloride decreased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 2
Blood culture positive (Investigations) | 0 | 1
Blood potassium decreased (Investigations) | 1 | 0
Breath sounds decreased (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchopneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chest discomfort (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Constipation (Gastrointestinal disorders) | 1 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 20 | 58
Crackles lung (Respiratory, thoracic and mediastinal disorders) | 1 | 7
Cyanosis (Cardiac disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 3 | 11
Dehydration (Metabolism and nutrition disorders) | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Distal intestinal obstruction syndrome (Gastrointestinal disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 | 30
Dyspnoea exacerbated (Respiratory, thoracic and mediastinal disorders) | 1 | 13
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1
Exercise tolerance decreased (General disorders) | 6 | 19
Fatigue (General disorders) | 4 | 10
Fluid retention (Renal and urinary disorders) | 0 | 1
Forced expiratory volume decreased (Investigations) | 1 | 3
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1
Gastrostomy tube insertion (Surgical and medical procedures) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 6 | 18
Headache (Nervous system disorders) | 2 | 4
Hepatitis acute (Hepatobiliary disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Increased viscosity of bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Infrequent bowel movements (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Lethargy (General disorders) | 0 | 3
Lipase increased (Investigations) | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Malaise (General disorders) | 1 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 2
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Non-cardiac chest pain (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Oxygen saturation decreased (Investigations) | 3 | 1
Oxygen supplementation (Surgical and medical procedures) | 1 | 1
Pain (General disorders) | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonia bacterial (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 12 | 46
Pulmonary function test decreased (Investigations) | 2 | 25
Pyrexia (General disorders) | 6 | 10
Rales (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 15
Respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Sputum purulent (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Urine output decreased (Investigations) | 0 | 1
Uterine leiomyoma (Reproductive system and breast disorders) | 0 | 1
Vocal cord paralysis (Nervous system disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 5
Weight decreased (Investigations) | 1 | 4
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 75 mg AZLI Two Times a Day (BID) (N=85) | 75 mg AZLI Three Times a Day (TID) (N=189)
Abdominal distension (Gastrointestinal disorders) | 4 | 11
Abdominal pain (Gastrointestinal disorders) | 10 | 20
Abdominal pain upper (Gastrointestinal disorders) | 12 | 20
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 | 25
Asthenia (General disorders) | 4 | 24
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 24
Blood glucose increased (Investigations) | 4 | 15
Breath sounds decreased (Respiratory, thoracic and mediastinal disorders) | 3 | 11
Chest discomfort (Respiratory, thoracic and mediastinal disorders) | 19 | 45
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 | 12
Chills (General disorders) | 7 | 19
Constipation (Gastrointestinal disorders) | 8 | 17
Cough (Respiratory, thoracic and mediastinal disorders) | 74 | 166
Crackles lung (Respiratory, thoracic and mediastinal disorders) | 26 | 37
Decreased appetite (Metabolism and nutrition disorders) | 25 | 83
Diarrhoea (Gastrointestinal disorders) | 10 | 30
Dizziness (Nervous system disorders) | 4 | 12
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 16
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 20 | 46
Dyspnoea exacerbated (Respiratory, thoracic and mediastinal disorders) | 6 | 25
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 7 | 22
Ear pain (Ear and labyrinth disorders) | 5 | 15
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 | 12
Exercise tolerance decreased (General disorders) | 42 | 104
Fatigue (General disorders) | 31 | 80
Forced expiratory volume decreased (Investigations) | 6 | 11
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 24 | 59
Headache (Nervous system disorders) | 25 | 61
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 12
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 17
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 33 | 70
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 7 | 10
Nasal oedema (Respiratory, thoracic and mediastinal disorders) | 9 | 5
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 2 | 10
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 7 | 5
Nausea (Gastrointestinal disorders) | 13 | 40
Non-cardiac chest pain (Respiratory, thoracic and mediastinal disorders) | 18 | 33
Pain (General disorders) | 8 | 17
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 15
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1 | 14
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 5 | 8
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 41 | 83
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 2 | 20
Productive cough (Respiratory, thoracic and mediastinal disorders) | 56 | 155
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 10
Pulmonary function test decreased (Investigations) | 10 | 37
Pyrexia (General disorders) | 38 | 83
Rales (Respiratory, thoracic and mediastinal disorders) | 5 | 6
Rash (Skin and subcutaneous tissue disorders) | 6 | 18
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 38 | 90
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 4 | 18
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 23 | 62
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 6 | 11
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 9 | 41
Sinus headache (Respiratory, thoracic and mediastinal disorders) | 9 | 30
Sneezing (Respiratory, thoracic and mediastinal disorders) | 3 | 14
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 1 | 19
Vomiting (Gastrointestinal disorders) | 18 | 38
Weight decreased (Investigations) | 13 | 24
Wheezing (Respiratory, thoracic and mediastinal disorders) | 26 | 50

LIMITATIONS AND CAVEATS:
Descriptive statistics for all participants receiving 1 or more doses of AZLI were summarized for the safety, microbiology, and efficacy endpoints. No formal hypothesis tests were planned. Rates of AEs and SAEs are not adjusted for time on study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution and investigator may publish or present the results of the trial generated there with prior written consent of Gilead; or 2 years after the trial has ended at all institutions. Proposed publications/target venue must go to Gilead 30 days (manuscripts) or 15 days (abstracts/presentations) prior. Any Gilead confidential information in the document(s) must be deleted or, if requested publication, delayed for up to 45 days to permit Gilead to obtain intellectual property protection.